CLINICAL TRIAL: NCT01712438
Title: Immunogenicity, Efficacy and Safety of Treatment With Human-cl-rhFVIII in Previously Untreated Patients With Severe Hemophilia A
Brief Title: Human Cell Line-derived Recombinant Factor VIII (Human-cl-rhFVIII) in Previously Untreated Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENA-05; 2012-002554-23 (EudraCT Number)
Record Dates: First submitted 2012-10-18; First posted 2012-10-23 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Severe Hemophilia A
Keywords: Previously untreated patients
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human cl rhFVIII (Experimental)
  Interventions: Biological: Human cl rhFVIII

INTERVENTIONS:
Biological: Human cl rhFVIII

SUMMARY:
Investigate the inhibitor development rate of Human cl rhFVIII in previously untreated patients with severe Hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Severe Hemophilia A (FVIII:C <1%)
* No previous treatment with FVIII concentrates or other blood products containing FVIII

Exclusion Criteria:

* Diagnosis with a coagulation disorder other than Hemophilia A
* Severe liver or kidney disease
* Concomitant treatment with any systemic immunosuppressive drug

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-02; Primary Completion 2018-12-14 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Knaub, Study Director — Octapharma
Locations (37):
- United States (3):
  - UC Davis, Sacramento, California
  - All Children's Hospital, St. Petersburg, Florida
  - Harvard Children's Hospital Boston, Boston, Massachusetts
- Republican Scientific Practical Center for Pediatric Oncology and Hematology, Minsk, Belarus
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Mc Master Children's Hospital, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Ste-Justine, Montreal, Quebec
- France (7):
  - L'hôpital Côte de Nacre - CHU de Caen, Caen
  - Centre de traitement de l'hemophilie, Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hopital de la Timone, Marseille
  - Hôtel-Dieu de Nantes, Centre Regional de Traitement de l'hemophilie, Nantes
  - Hôpital Necker, Paris
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Hopital Trousseau - CHU Tours, Tours
- Institute of Haematology and Transfusiology, Tbilisi, Georgia
- Germany (3):
  - Institut für Experimentelle Hämatologie und Transfusionsmedizin (IHT), Bonn
  - University Hospital Frankfurt/M, Frankfurt
  - Universitätsmedizin der Johannes-Gutenberg-Universität Mainz, Mainz
- India (3):
  - Kasturba Medical College, Dr. TMA Pai Hospital, Manipal, Karnataka
  - Sahyadri Speciality Hospital, Haematology & BMT Unit, Pune
  - Christian Medical College & Hospital, Dept of Haematology, Vellore
- Italy (2):
  - Univ. Di Perugia, Perugia
  - Centro di Referimento per le Malattie Emorragiche e Trombotiche, Torino
- Scientific Research Institute of Mother and Child Health Care, Chisinau, Moldova
- Centre Hospitalier Ibn Sina, Rabat, Morocco
- University Medical School Warsaw, Warsaw, Poland
- HSJ - Hospital de São João, EPE, Porto, Portugal
- Morozovsky Children's Hospital, Moscow, Russia
- Haemophilia Centre, University Clinical Centre, Ljubljana, Slovenia
- Spain (2):
  - Unitat d'hemofilia, Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
- Ukraine (2):
  - National Children's Specialized Hospital "OHMATDET", Kiev
  - Institute of Blood Pathology and Transfusion Medicine, Lviv
- United Kingdom (2):
  - Cambridge University Hospital, Cambridge
  - Great Ormond Street Hospital for Children, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Human-cl rhFVIII: Of the total number of patients that started in the study, the safety (SAF) and intent-to-treat (ITT) population received at least one treatment with Human-cl rhFVIII.
  Prophylactic treatment dose given to all patients in the PROPH population (all patients who received at least one administration of Human cI rhFVIII with prophylaxis documented as the reason for treatment): 20-50 IU/FVIII/kg body weight (BW)).
  On-demand treatment of bleeding episodes (BEs) dose given to the BLEED population (all patients with bleeding episodes treated with Human cI rhFVIII): 20-30 IU FVIII/kg BW (minor haemorrhage), 30-40 IU FVIII/kg BW (moderate to major haemorrhage) or 40-60 IU FVIII/kg BW (major to life-threatening haemorrhage). Surgical prophylaxis dose given to the SURG population (all patients with surgeries performed under Human cI rhFVIII treatment): 25-30 IU FVIII/kg BW (minor surgeries) or 40-60 IU FVIII/kg BW (major surgeries).
Period: Overall Study
Arm/Group | Human-cl rhFVIII
Started | 110
SAF Population (SAF population = study population of patients in safety analysis) | 108
ITT Population (ITT population = intent-to-treat population) | 108
PP Population (PP Population = per-protocol population) | 95
PROPH Population (PROPH population = study population of patients receiving prophylaxis) | 103
BLEED Population (BLEED population = study population of Bleeding Events (BEs)) | 94
SURG Population (SURG population = study population of patients undergoing surgery treated with Human-cl rhFVIII) | 24
Completed | 73
Not Completed | 37
Not completed — Not treated with Human-cl rhFVIII | 2
Not completed — Ongoing ITI treatment | 6
Not completed — Violated inclusion & exclusion criteria | 4
Not completed — Prematurely Discontinued | 25

BASELINE CHARACTERISTICS:
Population: The safety (SAF) and intent-to-treat (ITT) population consist of all patients who had data collected post-treatment with Human-cl rhFVIII (n=108).
Groups:
- Human-cl rhFVIII: The safety (SAF) and intent-to-treat (ITT) population consists all patients who had data collected post-treatment with Human-cl rhFVIII (n=108).
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 108
Age, Continuous [Mean (Full Range); unit: months] — Age at screening in months
  months | 19.0 [0 to 146]
Age, Continuous [Mean (Full Range); unit: months] — Age at exposure day 1 in months
  months | 21.6 [0 to 146]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 105
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 89
  More than one race | 0
  Unknown or Not Reported | 4
Body Mass Index (BMI) at Exposure Day 1 (ED1) [Mean (Full Range); unit: kg/m2] | 17.2 [9 to 43]
Height at Exposure Day 1 (ED1) [Mean (Full Range); unit: centimeters (cm)] — Height at exposure day 1 in centimeters
  centimeters (cm) | 82.0 [45 to 144]
Weight at Exposure Day 1 (ED1) [Mean (Full Range); unit: kilograms (kg)] — Weight at exposure day 1 in kilograms
  kilograms (kg) | 11.7 [3 to 31]
Family history of inhibitors [Count of Participants; unit: Participants]
  Yes | 13
  No | 95

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of Human-cl rhFVIII: Incidence of Inhibitors
Description: The number of patients developing FVIII inhibitors was observed during the observation period by assessing inhibitor development using the modified Bethesda assay (Nijmegen modification). The definitions for thresholds were ≥0.6 to <5 BU/mL for a "low titre" inhibitor and ≥5 BU/mL for a "high-titre" inhibitor.
Time Frame: maximum 5 years (100 exposure days)
Population: The analysis was performed for the SAF/ITT population which includes all patients who had data collected post-treatment with Human-cl rhFVIII (n=108). Of the 108 patients, 105 patients had at least one inhibitor test after exposure day (ED) 1.
Measure: Count of Participants; unit: Participants
Groups:
- SAF/ITT Population: All patients who had data collected post-treatment with Human-cl rhFVIII (n=108).
Arm/Group | SAF/ITT Population
Number analyzed (Participants) | 105
Participants
  High titre inhibitor (>5 BU/mL) | 17
  Low titre inhibitor (<5 BU/mL) | 11
  Any inhibitor (>0.6 BU/mL) | 28

2. Secondary Outcome: Frequency of Spontaneous Break-through Bleeds
Description: The annualized bleeding rate (ABR) was calculated during inhibitor-free periods for spontaneous bleeding events (BEs) during prophylactic treatment with Human cl rhFVIII
Time Frame: Maximum 5 years (100 exposure days)
Population: The analysis population includes all patients who received at least one prophylactic treatment with Human-cl rhFVIII (PROPH population; n=103). Of all patients in the PROPH population, data was available on spontaneous break-through bleeds for 102 patients.
Measure: Mean (95% Confidence Interval); unit: No. BEs per duration (year) (ABR)
Groups:
- PROPH Population: All patients who received at least one prophylactic treatment with Human-cl rhFVIII (n=103).
Arm/Group | PROPH Population
Number analyzed (Participants) | 102
No. BEs per duration (year) (ABR) | 0.976 [0.431 to 1.521]

3. Secondary Outcome: Efficacy of Human-cl rhFVIII for the Treatment of Bleeds
Description: A personal efficacy assessment to assess the efficacy of Human-cl rhFVIII for the on-demand treatment of bleeding episodes. Efficacy was assessed using a four-point scale (excellent, good, moderate, none).
Time Frame: Maximum 5 years (100 exposure days)
Population: The analysis population includes patients (n=94) who received Human-cl rhFVIII for on-demand treatment of BEs (BLEED population).
Measure: Count of Units; unit: Number of Bleeding Events
Units Other Than Participants: Number of Bleeding Events
Groups:
- BLEED Population: All patients that experienced at least one bleeding episode that was treated with Human-cl rhFVIII (n=94).
Arm/Group | BLEED Population
Number analyzed (Participants) | 94
Number analyzed (Number of Bleeding Events) | 804
Number of Bleeding Events
  Excellent | 510
  Good | 237
  Moderate | 51
  None | 6

4. Secondary Outcome: Efficacy of Human-cl rhFVIII for Surgical Prophylaxis
Description: An overall efficacy assessment to assess the efficacy of human-cl rhFVIII in surgical prophylaxis of minor and major surgeries. The efficacy assessment was analyzed using a four-point scale (excellent, good, moderate, none).
Time Frame: Maximum 5 years (100 exposure days)
Population: The analysis population includes 24 patients that received Human-cl rhFVIII for surgical prophylaxis during a total of 26 surgeries (SURG population). Of these, 13 patients had minor surgeries and 11 patients had major surgeries. Of the total 26 surgeries, 21 had an overall efficacy assessment (an assessment was not performed for 5 surgeries).
Measure: Count of Units; unit: Number of surgeries
Units Other Than Participants: Number of surgeries
Groups:
- Minor Surgeries: All patients that had minor surgeries performed under Human-cl rhFVIII treatment (n=13)
- Major Surgeries: All patients that had major surgeries performed under Human-cl rhFVIII treatment (n=11)
- All Surgeries: All patients that had surgeries performed under Human-cl rhFVIII treatment (n=24)
Arm/Group | Minor Surgeries | Major Surgeries | All Surgeries
Number analyzed (Participants) | 13 | 11 | 24
Number analyzed (Number of surgeries) | 10 | 11 | 21
Number of surgeries
  Excellent | 7 | 8 | 15
  Good | 1 | 2 | 3
  Moderate | 1 | 1 | 2
  None | 1 | 0 | 1

5. Other Pre Specified Outcome: The Occurrence of Any Adverse Event (AE)
Description: The frequency of AEs, as monitored throughout the whole study by the number of patients with at least one adverse event occurrence.
Time Frame: 5 years
Population: Of the 110 patients enrolled in the study, 2 were excluded because they had no treatment with Human-cl rhFVIII leaving 108 patients in the safety (SAF) and intent-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | SAF/ITT Population
Number analyzed (Participants) | 108
Participants
  Adverse Event (AE) | 101
  Serious adverse event (SAE) | 48
  Severe AE | 27
  Temporally related adverse event | 78
  Death | 0
  Death due to probably/possibly related AE | 0
  AE leading to permanent study discontinuation | 2

ADVERSE EVENTS:
Time Frame: Maximum 5 years (100 exposure days)
Arm/Group | SAF/ITT Population
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 48/108
Other Adverse Events (participants affected / at risk) | 101/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAF/ITT Population (N=108)
Factor VIII inhibition (Blood and lymphatic system disorders) | 28 (29)
Haematoma (Vascular disorders) | 4 (4)
Tonsillitis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 5 (8)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Device Issue (Product Issues) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Factor IX inhibition (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2)
Device related sepsis (Infections and infestations) | 2 (3)
Device related infection (Infections and infestations) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAF/ITT Population (N=108)
Nasopharyngitis (Infections and infestations) | 35
Rhinitis (Infections and infestations) | 20
Upper respiratory tract infection (Infections and infestations) | 12
Ear infection (Infections and infestations) | 11
Bronchitis (Infections and infestations) | 10
Conjunctivitis (Infections and infestations) | 9
Gastroenteritis (Infections and infestations) | 9
Varicella (Infections and infestations) | 8
Respiratory tract infection (Infections and infestations) | 7
Laryngitis (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 5
Tonsillitis (Infections and infestations) | 5
Lower respiratory tract infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Device related information (Infections and infestations) | 3
Erythema infectiosum (Infections and infestations) | 3
Influenza (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Pyrexia (General disorders) | 61
Factor VIII inhibition (Blood and lymphatic system disorders) | 28
Anaemia (Blood and lymphatic system disorders) | 21
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 14
Teething (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 12
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Head injury (Injury, poisoning and procedural complications) | 6
Mouth injury (Injury, poisoning and procedural complications) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Haemoglobin decreased (Investigations) | 4
Iron deficiency (Metabolism and nutrition disorders) | 4
Hypersensitivity (Immune system disorders) | 3
Haematoma (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT01712438/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT01712438/SAP_003.pdf